CLINICAL TRIAL: NCT02018419
Title: In-Situ Cancer Vaccine: Phase I/IIb, Open-Label Study to Assess Safety of AllostimTM in Combination With Cryoablation in Metastatic Breast Cancer Previously Treated With an Anthracycline, a Taxane and Capecitabine
Brief Title: Increased Frequency of AlloStim(TM) Dosing in Combination With Cryoablation in Metastatic Breast Cancer Patients
Acronym: MBC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: changing indication from breast cancer to metastatic colorectal cancer
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-014-TACT-MBC
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2015-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Schedule A (Experimental): 1. the priming step with ID injection of AlloStim on Days 0, 7, and 14;
  2. the ablation step with cryoablation and intra-tumor injection of AlloStim on Day 21;
  3. the activation step with an IV infusion of AlloStim on Day 28;
  4. the booster step with intravenous booster infusion of AlloStim on Days 56 and 84;
  Protocol follow-up procedures continue until day 168 and at investigator discretion thereafter.
  Interventions: Biological: AlloStim; Procedure: Cryoablation
- Dosing Schedule B (Experimental): 1. the priming step with ID injection of AlloStim on Days 0 and 3 and an additional ID injection of AlloStim on Days 7 and 10;
  2. the ablation step with cryoablation and intra-tumor injection of AlloStim on Day 14;
  3. the activation step with an IV infusion of AlloStim on Day 21;
  4. the booster step with intravenous booster infusion of AlloStim on Days 49 and 77.
  Protocol follow-up procedures continue until day 168 and at investigator discretion thereafter.
  Interventions: Biological: AlloStim; Procedure: Cryoablation
- Dosing Schedule C (Experimental): 1. the priming step with ID injection of AlloStim on Days 0 and 3 and an additional ID injection of AlloStim on Days 7 and 10;
  2. the ablation step with cryoablation and intra-tumor injection of AlloStim on Day 14, and intra-tumor injection of AlloStim again into the same cryoablated lesion on Day 17;
  3. the activation step with an IV infusion of AlloStim on Day 21;
  4. the booster step with intravenous infusion of AlloStim on days 49 and 77.
  Protocol follow-up procedures continue until day 168 and at investigator discretion thereafter.
  Interventions: Biological: AlloStim; Procedure: Cryoablation

INTERVENTIONS:
Biological: AlloStim — AlloStim is derived from the blood of normal blood donors and is intentionally mismatched to the recipient.
  Other Names: InSituVax; Personalized anti-tumor vaccine
Procedure: Cryoablation — Percutaneous ablation of a single metastatic tumor lesion usually in liver or bone. The procedure is conducted under CT or ultrasound image-guidance.

SUMMARY:
This phase I/II study is designed to compare different treatment schedules of a personalized anti-cancer vaccine protocol which combines the cryoablation of a selected metastatic lesion with intra-tumor immunotherapy. The cryoablation causes the tumor to release tumor-specific antigens into the surrounding environment. The injection of bioengineered allogeneic immune cells, AlloStim(TM), into the lesion is designed to modulate the immune response and educate the immune system to kill other tumor cells.

DETAILED DESCRIPTION:
The study will assess three different dosing schedules. A standard 3 plus 3 study design will be used. The starting dose for each dosing schedule will be escalated in subsequent groups of patients. The study will evaluate safety of increased frequency of AlloStim (TM) dosing and anti-tumor effect of the new proposed dose and frequency schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Women w/ histologically/cytologically confirmed breast carcinoma
2. Documented progressive metastatic disease not amenable to curative surgery/radiotherapy
3. Age ≥18 and ≤70 years
4. Prior treatments that included capecitabine and both an anthracycline and a taxane drug and resistant to taxane therapy

   1. ER+ patients: minimum cumulative dose of anthracycline (≥ 180 mg/m² of doxorubicin or ≥ 300 mg/m² of epirubicin) or resistance to anthracycline, capecitabine and anti-hormonal therapy
   2. Resistance is defined as tumor progression while receiving treatment or progression within 4 months of the last dose in the metastatic setting, or recurrence within 12 months in the neoadjuvant/adjuvant setting
5. Post-menopausal ER+ and/or PR+ must have received at least 2 lines of prior anti-estrogen therapy, which includes an aromatase inhibitor
6. Her2+ patients: at least 1 Her2+ targeted regimen containing trastuzumab alone or with pertuzumab/lapatinib. Trastuzumab/pertuzumab must have been discontinued at least 4 weeks before treatment
7. Prior radiation therapy completed >4 weeks before treatment
8. Measurable disease according to revised RECIST v.1.1 guidelines with at least 1 lesion deemed to be safely accessible for serial biopsy
9. ECOG <2
10. Adequate hematological function

    1. Absolute granulocyte count ≥ 1,500/mm3
    2. Platelet count ≥ 100,000/mm3
    3. PT/INR ≤ 1.5
    4. INR correctable to ≤ 1.5 or a PT/PTT correctable to normal limits. Patients receiving anti-coagulation treatment with agent such as warfarin/heparin may participate. For patients on warfarin, INR should be monitored weekly prior to any intervention to assure INR is stable. Heparin/warfarin must be withheld before biopsy
    5. Hemoglobin ≥ 9 g/dL (may be corrected by transfusion)
11. Adequate organ function

    1. Creatinine ≤ 1.5 mg/dL
    2. Total bilirubin ≤ 1.5 times ULN
    3. Alkaline phosphatase≤2.5 times ULN (≤5 times normal if liver involvement)
    4. Aspartate aminotransferase (AST/SGOT) ≤ 5.0 times ULN
    5. Alanine aminotransferase (ALT/SGPT) ≤ 5.0 times ULN
12. EKG without clinically relevant abnormalities
13. Pre-menopausal with child bearing potential subjects must use adequate contraception
14. Informed consent in the native language of the subject

Exclusion Criteria:

1. Peritoneal carcinomatosis
2. Moderate-large ascites accumulation requiring/likely to require paracentesis
3. Clinical/radiological evidence of brain metastasis/leptomeningeal involvement
4. Pulmonary lymphangitis/symptomatic pleural effusion (grade ≥ 2) that results in pulmonary dysfunction requiring active treatment
5. History of 2nd primary malignancy, except: bilateral breast carcinoma, in situ carcinoma of the cervix, adequately treated non-melanomatous carcinoma of the skin, and other malignancy treated at least 5 years with no evidence of recurrence
6. >3 prior chemotherapy regimens for metastatic disease
7. History of severe hypersensitivity to monoclonal antibody drugs/any contraindication to study drugs
8. Pregnant or breast feeding
9. Any serious, concurrent uncontrolled medical disorder
10. Prior hepatectomy, liver chemoembolization, liver cryoablation/ radiofrequency ablated
11. Symptomatic pulmonary disease
12. Bevacizumab (Avastin®) within 3 weeks of accrual
13. Prior allogeneic bone marrow/stem cell or solid organ transplant
14. Chronic use (> 2 weeks) of greater than physiologic doses of corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 30 days of the first day of study treatment. Topical and inhaled corticosteroids are permitted
15. Concomitant active autoimmune disease
16. Prior experimental therapy/cancer vaccine treatment
17. Current immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 1 month of study entry
18. History of blood transfusion reactions
19. Known allergy to bovine products
20. Know allergy to murine products
21. Progressive viral/bacterial infection. All infections must be resolved and the patient must remain afebrile for 7days without antibiotics prior to enrollment
22. Cardiac disease of symptomatic nature or cardiac ejection fraction < 45%
23. History of HIV positivity or AIDS
24. Psychiatric/addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation
25. Concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to cryoablation procedure
26. Use of low molecular weight heparin preparations unless can be discontinued 8 hours prior to cryoablation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety of increased frequency of dosing | Window is defined as the time required receiving two doses of AlloStim IV push plus 28 days follow-up
  Three patients are enrolled at each frequency schedule in the absence of dose limiting toxicity (DLT). A DLT is defined as any allergic or autoimmune toxicity or other study drug related toxicity Grade 3 or higher during the DLT assessment window.

SECONDARY OUTCOMES:
Health-Related Quality of Life | From enrollment to 90 days after last dose administration.
  Health-Related Quality of life will be measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) and its supplementary breast cancer questionnaire (QLQ-BR23).
Evaluate the anti-tumor effect of Allostim combined with cryoablation at the new proposed dose and frequency schedule. | 90 days after last dose administration
  Each treatment schedule will be monitored for radiological, pathological, and immunological response. These assessments will be compared between three treatment schedules.

OTHER OUTCOMES:
Immunological Response | 90 days after last dose administration
  Blood samples will be evaluated for immunological response and a determination made as to whether immunological response correlates with RECIST and pathology.
Anti-Tumor Response | 90 days after last dose administration
  The changes in tumor burden by RECIST and compare these changes with the pathological analysis of corresponding biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Zivile Katiliene, Ph.D., Study Director — Immunovative Clinical Research
Locations (1):
- Medical Oncology Associates of San Diego, San Diego, California, United States

REFERENCES:
- [Result] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441
- [Result] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Result] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Result] Janikashvili N, LaCasse CJ, Larmonier C, Trad M, Herrell A, Bustamante S, Bonnotte B, Har-Noy M, Larmonier N, Katsanis E. Allogeneic effector/memory Th-1 cells impair FoxP3+ regulatory T lymphocytes and synergize with chaperone-rich cell lysate vaccine to treat leukemia. Blood. 2011 Feb 3;117(5):1555-64. doi: 10.1182/blood-2010-06-288621. Epub 2010 Dec 1. PMID 21123824
- [Result] LaCasse CJ, Janikashvili N, Larmonier CB, Alizadeh D, Hanke N, Kartchner J, Situ E, Centuori S, Har-Noy M, Bonnotte B, Katsanis E, Larmonier N. Th-1 lymphocytes induce dendritic cell tumor killing activity by an IFN-gamma-dependent mechanism. J Immunol. 2011 Dec 15;187(12):6310-7. doi: 10.4049/jimmunol.1101812. Epub 2011 Nov 9. PMID 22075702